CLINICAL TRIAL: NCT06299748
Title: A Worldwide Pregnancy Safety Study To Assess Maternal, Fetal, And Infant Outcomes Following Exposure To Efgartigimod During Pregnancy And/Or Breastfeeding
Status: Recruiting | Type: Observational
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Other Study IDs: ARGX-113-PAC-2206
Record Dates: First submitted 2024-02-22; First posted 2024-03-08 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Myasthenia Gravis; CIDP - Chronic Inflammatory Demyelinating Polyneuropathy
MeSH Terms: conditions — Myasthenia Gravis; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — efgartigimod alfa

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective Pregnancy: woman is no longer pregnant at time of study enrollment but was exposed to efgartigimod or efgartigimod PH20 SC any time within 25 days prior to conception or any time during pregnancy
  Interventions: Biological: Efgartigimod
- Prospective Pregnancy: woman is pregnant or breastfeeding at time of study enrollment.
  Interventions: Biological: Efgartigimod

INTERVENTIONS:
Biological: Efgartigimod — Efgartigimod IV or SC

SUMMARY:
This is a multi-country, prospective safety study of pregnant women exposed to efgartigimod or efgartigimod PH20 SC any time within 25 days prior to conception or any time during pregnancy. Women exposed to efgartigimod or efgartigimod PH20 SC only during breastfeeding will also be eligible to enroll. Background rates of major congenital malformations (MCMs) will be obtained from populations within the same countries/regions as the countries/regions in which the efgartigimod or efgartigimod PH20 SC exposed pregnancies were reported.

ELIGIBILITY:
Inclusion Criteria:

* Women with exposure to efgartigimod or efgartigimod PH20 SC any time within 25 days prior to conception or any time during pregnancy, or women with exposure to efgartigimod or efgartigimod PH20 SC during breastfeeding. The timeframe of 25 days prior to conception is calculated based on five times the efgartigimod half-life, which is 3 to 5 days.
* Written/verbal informed consent or eConsent (depending on country regulations) (for adolescents under the age of majority, written/verbal informed assent or eConsent by the pregnant minor (where applicable) and written/verbal informed consent or eConsent by the parent/legal guardian).

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women or women no longer pregnant at the time of study enrollment but exposed to efgartigimod any time within 25 days prior to conception or any time during the pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 279 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2033-01 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Pregnancy outcomes | up to 10 years
  Pregnancy outcomes: Spontaneous abortion; Elective or therapeutic abortion; Fetal death/stillbirth ; Molar or ectopic pregnancy; Live birth (Preterm delivery; Fullterm delivery)

SECONDARY OUTCOMES:
Congenital malformations | up to 10 years
  Congenital malformations (CDC 2020b) identified in the developing fetus, neonate, or infant: Major congenital malformations (MCMs); Minor congenital malformations
The number of observed other events of interest in the developing neonate and infant (such as hospitalizations for serious illness) | up to 10 years
  Other events of interest identified in the developing neonate and infant (Hospitalizations for serious illness; Potential adverse reactions to medications; Growth and development milestones as described by the Centers for Disease Control and Prevention or other accepted standard assessments; Infant developmental deficiency; Postnatal growth deficiency or failure to thrive (FTT); Neonatal and infant mortality; Infections; Transient neonatal myasthenia; Vaccination and vaccine reactions
Maternal complications of pregnancy | up to 10 years
  Maternal complications of pregnancy, including but not limited to: Premature rupture of membranes (PROM); Preterm PROM (PPROM); Pre-eclampsia; Gestational hypertension; Eclampsia; Proteinuria; Gestational diabetes; Intrauterine growth restriction (IUGR); Polyhdramnios
Maternal infections | up to 10 years
The number of observed fetal growth deficiency | up to 10 years

CONTACTS AND LOCATIONS:
Locations (4):
- United BioSource LLC, Morgantown, West Virginia, United States
- Klinikum der Ruhr-Universität Bochum St. Josef Hospital Neurologische Interdisziplinäre Infusionsambulanz + MS Studienambulanz (Haus E Ebene1), Bochum, Germany
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided